CLINICAL TRIAL: NCT06503822
Title: Comparison of Application Effects Between Long Peripheral Venous Catheters and Standard Short Peripheral Venous Catheters: A Multicenter Prospective Randomized Controlled Trial Study
Brief Title: Comparison of Application Effects Between Long- and Standard Short- Peripheral Venous Catheters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Third People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-089-02
Record Dates: First submitted 2024-06-27; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Hospitalized Patients
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In the intervention group, a new long peripheral venous catheter was selected by the puncture operator according to the puncture location and venous conditions, and was placed using aseptic technology. After blood return, the catheter could be easily rinsed with 0.9% sodium chloride solution, which was considered to be placed in the correct position and could be used normally. Intravenous infusion therapy begins immediately after successful catheterization. Check the condition of the catheter at least 3 times a day, and rinse with 10 ml.9% sodium chloride solution before each intravenous treatment; After disconnection of any infusion, pulse flushing with 0.9% sodium chloride solution 10ml and positive pressure sealing tube flushing to seal the catheter. Collect patient information, including sociodemographic information, duration of intravenous therapy, and details about catheter failure.
  Interventions: Device: Long peripheral venous catheter
- Control group (Active Comparator): The control group will receive a new 24G or 22G short peripheral venous catheter with direct view aseptic technique puncture, see blood return and rinse easily with 0.9% sodium chloride solution. The catheter is considered to be in the correct position and can be used normally. Check the condition of the catheter at least 3 times a day, and rinse with 10 ml.9% sodium chloride solution before each intravenous treatment; After disconnection of any infusion, pulse flushing with 0.9% sodium chloride solution 10ml and positive pressure sealing tube flushing to seal the catheter. Collect patient information, including sociodemographic information, duration of intravenous therapy, and details about catheter failure.
  Interventions: Other: Control group (Short peripheral venous catheter)

INTERVENTIONS:
Device: Long peripheral venous catheter — In this study, patients eligible for admission were subjected to peripheral vein long catheter puncture according to the operating standards, daily routine maintenance until catheter removal, and relevant data were collected.
  Arms: Intervention group
Other: Control group (Short peripheral venous catheter) — In this study, the patients eligible for admission will undergo peripheral venous short catheter puncture according to the operating standards, daily routine maintenance until catheter removal, and relevant data will be collected.
  Other Names: Short peripheral venous catheter
  Arms: Control group

SUMMARY:
Short PIVC (intravenous indentation needle) accounts for more than 50% of clinical infusion tools, but long PIVC is rarely used and studied in China. This study aims to explore the application characteristics and application effects of long PIVC in China. It provides reference for the correct selection of infusion tools, and promotes the clinical application and promotion of new intravenous therapy tools.

The study nurse will work with the responsible physician to assess the eligibility for enrollment and sign the informed consent. Were randomly assigned to the control group (to receive a new 24G/22G (0.7mm*19mm/0.9mm*25mm) short PIVC (closed needle protected venous catheter system) puncture) or the intervention group (to insert a new 3F (8cm) or 4F(10cm) long PIVC) for daily routine maintenance until catheter removal, General demographic data, laboratory-related data, catheter-related data, catheter-related complications (unplanned extubation, phlebitis, catheter blockage, catheter-related thrombosis, catheter-related bloodstream infection, exudation, etc.) and patient satisfaction were collected.

DETAILED DESCRIPTION:
The control group will receive a new 24G or 22G short peripheral venous catheter for puncture using direct view aseptic technique, while the intervention group will be implanted with a new long peripheral venous catheter selected by the puncture operator using aseptic technique depending on the puncture location and venous conditions. After successful puncture, blood was returned in both groups and easily washed with 0.9% sodium chloride solution. The catheter was considered to be placed in the correct position and could be used normally. Intravenous infusion therapy should be started immediately after successful catheterization. The catheter should be checked at least 3 times a day and washed with 10 ml.9% sodium chloride solution before each intravenous therapy. After disconnection of any infusion, pulse flushing with 0.9% sodium chloride solution 10ml and positive pressure sealing tube flushing to seal the catheter. Patient information was collected during the study, including sociodemographic information, duration of intravenous therapy, and details about catheter failure.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female aged 18 years or older who is able and willing to give written informed consent;
2. Identification of the patient's medical diagnosis based on the competent physician and the study nurse at any time during the hospital stay, and judgment that the duration of peripheral intravenous infusion therapy needs to exceed 4 days;
3. Subjects with good compliance and can cooperate with catheter maintenance and observation.

Exclusion Criteria:

1. Patients who are delirious and unable to cooperate;
2. Patients requiring central venous access;
3. Patients suffering from connective tissue diseases or blood diseases;
4. Patients allergic to catheters or dressings;
5. any subject in a condition deemed by the investigator to interfere with the evaluation of results or pose a health risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Unplanned extubation | Up to 2 months
  Any complications of catheter removal before completion of IV therapy or before the recommended time of catheter use. Removal of the catheter at the end of intravenous infusion therapy is not considered catheter failure.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoning Liu, Study Chair — Shenzhen Third People's Hospital
Locations (1):
- Deng Qiuxia, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No